CLINICAL TRIAL: NCT01366092
Title: A Phase II Trial of Daily Low-Dose Interleukin-2 (IL-2) for Steroid-Refractory Chronic Graft-Versus-Host-Disease
Brief Title: Daily IL-2 for Steroid-Refractory Chronic Graft-versus-Host-Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Prometheus Laboratories (Industry)
Responsible Party: Principal Investigator, John Koreth, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-149; P01CA142106 (NIH)
Record Dates: First submitted 2011-06-02; First posted 2011-06-03 (Estimated); Results first posted 2015-01-15 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Chronic Graft-versus-host Disease
Keywords: stem cell transplant; GVHD; bone marrow transplant; cord blood transplant; regulatory T cell; interleukin
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interleukin-2 (Experimental): Each study participant will receive daily subcutaneous IL-2 (1 x 106 IU/m2/day) for self-administration for 12 weeks, followed by a 4-week hiatus. IL-2 will be typically administered on an outpatient basis. After completing the 16 week study (12 weeks of IL-2 study treatment and a mandatory 4 weeks off-IL-2), patients experiencing clinical benefit (complete or partial response; as well as minor response not meeting NIH criteria for partial response) with an acceptable toxicity profile will be permitted to continue extended-duration treatment indefinitely at the discretion of the treating physician.
  Interventions: Drug: Interleukin-2

INTERVENTIONS:
Drug: Interleukin-2 — Daily subcutaneous IL-2 (1 x 10^6 IU/m^2/day) for self-administration for 12 weeks followed by 4-week hiatus
  Other Names: IL-2

SUMMARY:
Chronic GVHD is a medical condition that may occur after a bone marrow, stem cell or cord blood transplant. The donor's immune system may recognize the your body (the host) as foreign and attempt to 'reject' it. This process is known as graft-versus-host-disease. It is thought that IL-2 may help control chronic GVHD by stopping the donor's immune system from 'rejecting' your body. In this research study, we are looking to see how IL-2 can be used in combination with steroids to treat cGVHD.

DETAILED DESCRIPTION:
You will give yourself or be given IL-2 daily through an injection under your skin. You should rotate the injection site, if possible. You will do this once every day for 12 weeks. You will then have 4 weeks off of IL-2. During the first 6 weeks of IL-2, you will continue to take steroids without changing the dose your doctor has set for you while you are on IL-2. After 6 weeks of IL-2 therapy, your doctor may reduce the amount of steroids you take.

While you are on study, a member of the study team will examine you to evaluate your cGVHD. These assessments may include examination of your skin, joints/muscles, eyes, mouth, lungs and gastrointestinal system.

You will have clinic visits for evaluation of toxicity and clinical benefit approximately every 4 weeks. You will also have immunologic assays approximately every 8 weeks. Immunologic assays will measure the effect of IL-2 on immune cells.

You will be on the study for about 16 weeks. You may continue on study treatment for longer if you experience a clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of allogeneic stem cell transplantation with myeloablative or non-myeloablative conditioning regimens
* Steroid refractory cGVHD with systemic therapy onset within the prior 6 months
* No more than 2 prior lines of cGVHD therapy
* Estimated life expectancy > 3 months
* Adequate organ function

Exclusion Criteria:

* Ongoing prednisone requirement > 1 mg/kg/day (or equivalent)
* Concurrent use of calcineurin-inhibitors plus sirolimus
* History of thrombotic microangiopathy, hemolytic-uremic syndrome or thrombotic thrombocytopenic purpura
* Active malignant relapse
* Active uncontrolled infection
* Uncontrolled cardiac angina or symptomatic congestive heart failure
* Organ transplant (allograft) recipient
* HIV-positive on combination antiretroviral therapy
* Active hepatitis B or C
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-07; Primary Completion 2014-10 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John Koreth, MBBS, DPhil, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Interleukin-2
Started | 35
Completed | 31
Not Completed | 4
Not completed — Progressive cGVHD | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Interleukin-2
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 51 [22 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 35
Time from Allogeneic Stem Cell Transplant [Median (Full Range); unit: days] | 616 [270 to 2145]
Time from chronic GVHD onsent [Median (Full Range); unit: days] | 252 [28 to 1880]
Number of cGVHD organ sites [Median (Full Range); unit: organs affected by cGVHD] | 4 [1 to 7]
Number of concurrent cGVHD therapies [Median (Full Range); unit: therapies] | 2 [1 to 3]
Baseline Corticosteroid (Prednisone) dose [Median (Full Range); unit: milligrams per day] | 20 [2.5 to 50]

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate of Low-dose Daily SC IL-2 in Steroid-refractory cGVHD
Description: Participants were evaluated according to the cGVHD NIH Consensus criteria at baseline, 6 weeks, and 12 weeks on study. Per cGVHD NIH Consensus criteria, cGVHD involved organ systems are given a grade 0-3 and an overall cGVHD score, from 0-10, is given. Complete Response is defined as resolution of all reversible manifestations in each organ or site of cGVHD. A partial response is defined as an improvement in measure at least one organ or site, or decrease in global ratings by at least a 2-point change on the 10-point scale, without progression measured at any other organ or site. Non-responders have no change in cGVHD meeting criteria for either partial response or disease progression. Progressive disease is defined as an increase in organ or site scales (1-point change on a 3-point scale) or 2- to 3-point increase on the global cGVHD ratings. Clinical worsening of cGVHD is not synonymous with progressive cGVHD per NIH criteria.
Time Frame: Baseline, 6 weeks, and 12 weeks
Population: 33 of 35 patients were evaluable for response criteria. To be evaluable, patients had to receive at least 6 weeks of daily IL-2 and had their disease re-assessed.
Measure: Number; unit: participants
Arm/Group | Interleukin-2
Number analyzed (Participants) | 33
participants
  Overall Partial Response | 21
  Overall Stable Response | 10
  Overall cGVHD Progression | 2
  Skin cGVHD Response | 9
  Joint/Fascia/Muscle cGVHD Response | 4
  Liver cGVHD Response | 7
  Lung cGVHD Response | 3
  GI tract cGVHD Response | 4

2. Secondary Outcome: Toxicity of 12-week Course of Low-dose SC IL-2 Therapy
Description: Participants were evaluated at clinical visits for toxicities related to IL-2 throughout their 12-week treatment course
Time Frame: 12 weeks
Population: Grade 2 or higher, related to IL-2, adverse events (AE) were recorded for participants during their 12-week IL-2 treatment course. AE's were evaluated based on the CTCAE version 4.0.
Measure: Number; unit: Grade 2 or higher related AEs
Arm/Group | Interleukin-2
Number analyzed (Participants) | 35
Grade 2 or higher related AEs | 3

3. Secondary Outcome: Prednisone Taper With IL-2 Therapy
Description: Participants had their steroid dose assessed at weeks 6, 12,16, and every 8 weeks while on extended duration IL-2 therapy.
Time Frame: End of treatment after 16 weeks or most recent follow-up date for patients on extended
Population: Participant's steroid taper was measured using their steroid dose at the start of therapy and their dose at the end of 16 weeks. For participants who continued on extended duration therapy, their final steroid dose was determined at the time of stopping treatment or, if still ongoing, the last clinic visit at the time of data analysis.
Measure: Mean (Full Range); unit: percent taper
Arm/Group | Interleukin-2
Number analyzed (Participants) | 33
percent taper | 42.8 [0 to 100]

4. Secondary Outcome: Overall Survival and Progression-free Survival
Description: Overall survival (OS) and progression-free survival (PFS) were calculated using the Kaplan-Meier method. OS was defined as from the study entry to death from any cause. Patients who were alive or lost to follow-up were censored at the time last seen alive. PFS was defined from the study entry to disease relapse or progression or death from any cause, whichever occurred first.
Time Frame: 2 years from start of IL-2
Measure: Number; unit: probability
Arm/Group | Interleukin-2
Number analyzed (Participants) | 33
probability
  Overall Survival | 0.91
  Progression-Free Survival | 0.82

5. Secondary Outcome: Immunologic Effects of Low-dose Daily SC IL-2: Treg Cell Counts
Description: Blood samples were collected throughout the patient's 12 weeks of IL-2 treatment and after the 4 week hiatus. The CD4+CD25+FOXP3+ regulatory T cells (Treg) counts were measured.
Time Frame: 16 weeks of study follow-up
Measure: Median (Inter-Quartile Range); unit: cell count/ uL
Arm/Group | Interleukin-2
Number analyzed (Participants) | 35
cell count/ uL
  Baseline regulatory T cell | 17.1 [8.6 to 40.6]
  Week 4 Treg cell count | 137.9 [51.8 to 188]
  Week 12 Treg cell count | 104.1 [53.9 to 167.1]

6. Secondary Outcome: Immunologic Effects of Low-dose Daily SC IL-2: Treg/Tcon Ratio
Description: Blood samples were collected throughout the patient's 12 weeks of IL-2 treatment and after the 4 week hiatus. The ratio between CD4+CD25+FOXP3+ regulatory T cells (Treg) and CD4 conventional T cell (Tcon) counts were measured.
Time Frame: 16 weeks of study follow-up
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Interleukin-2
Number analyzed (Participants) | 35
ratio
  Baseline Treg:Tcon ratio | 0.06 [0.05 to 0.13]
  Week 2 Treg:Tcon ratio | 0.35 [0.26 to 0.48]
  Week 12 Treg:Tcon ratio | 0.31 [0.27 to 0.39]

ADVERSE EVENTS:
Time Frame: From first dose of study drug at Week 1 until Week 16 visit.
Description: Participants were evaluated for adverse events at every clinical visit during Weeks 1,2,4,6,8.10,12,16 and every 4 weeks on extended duration therapy. Only serious adverse events and other adverse events that occurred during the 16-week study period are recorded here. Per protocol, only AEs Grade 3 or higher were recorded.
Arm/Group | Interleukin-2
Serious Adverse Events (participants affected / at risk) | 4/35
Other Adverse Events (participants affected / at risk) | 10/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interleukin-2 (N=35)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3) — These events were deemed unrelated to study treatment
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) — These events were deemed unrelated to study treatment
Streptococcus viridans infection (Infections and infestations) | 1 (1) — This event was deemed unrelated to study treatment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interleukin-2 (N=35)
Platelet count decreased (Blood and lymphatic system disorders) | 1 (1) — This event was deemed possibly related to study treatment
Fatigue (General disorders) | 1 (1) — This event was deemed probably related to study treatment
Flu-like symptoms (General disorders) | 1 (1) — This event was deemed related to study treatment
Hypertension (Cardiac disorders) | 2 (3) — This event was deemed unrelated to study therapy
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) — This event was deemed unrelated to study therapy
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) — This event was deemed unrelated to study therapy
Peripheral Motor Neuropathy (Nervous system disorders) | 1 (1) — This event was deemed unrelated to study therapy
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (4) — This event was deemed unrelated to study therapy
Thromoembolic Event (Vascular disorders) | 2 (2) — This event was deemed unrelated to study therapy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No